CLINICAL TRIAL: NCT06745869
Title: Effects of Aerobic and Diaphragmatic Breathing Exercises on Respiratory Functions and Voice Performance of Choir Singers
Brief Title: Effects of Aerobic and Diaphragmatic Exercises on Choir Singers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Sıla YILMAZ, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-197
Record Dates: First submitted 2024-12-10; First posted 2024-12-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Muscles; Cardiorespiratory Fitness
Keywords: Singing; Respiratory Function Tests; Voice; Diaphragm; Exercise, aerobic
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The researcher who evaluated the analysis, and the participants are blind to the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- diaphragmatic breathing exercise training group (Active Comparator): Participants included in the diaphragmatic breathing exercise training group will be provided diaphragmatic breathing training by a physiotherapist before starting the exercise program.
  Interventions: Behavioral: Diaphragmatic breathing exercise training
- aerobic exercise training group (Experimental): The protocol given to the diaphragmatic breathing exercise training group will also be included in the exercise program of participants included in the aerobic exercise training group.
  Interventions: Behavioral: Diaphragmatic breathing exercise training; Behavioral: Aerobic exercise training
- Control group (No Intervention): Participants included in the control group will be asked to continue their daily routines without changing their lifestyles.

INTERVENTIONS:
Behavioral: Diaphragmatic breathing exercise training — At the end of the training, participants will be asked to do an exercise session and this session will be observed. Training will continue until participants learn and apply the exercise correctly.
  5-minute warm-up and cool-down periods will be applied at the beginning and end of each exercise session. Exercises will be done twice a day, morning and evening, for 8 weeks.
  In order to follow the exercise, participants will be given diaphragmatic breathing exercise tracking cards with date and session information. In addition, participants will be followed up weekly on one of the rehearsal days to ensure their adaptation to the exercise.
  Arms: aerobic exercise training group; diaphragmatic breathing exercise training group
Behavioral: Aerobic exercise training — The intensity of the aerobic exercise program will be calculated for each participant using the Karvonen formula. Accordingly, each participant will be given a brisk walking program on a suitable surface, which will be created specifically for the individual to reach the target heart rate range within the scope of the aerobic exercise program; they will apply a 45-minute session, 3 days a week, for 8 weeks.
  Arms: aerobic exercise training group

SUMMARY:
The goal of this randomized-controlled study is to compare the effects of diaphragmatic breathing exercise training provided by a physiotherapist and aerobic exercise training applied in addition to diaphragmatic breathing exercise training provided by a physiotherapist on respiratory functions and voice performance in choir singers.

The main questions this study aims to answer are:

* Is diaphragmatic breathing exercise training provided by a physiotherapist effective in improving the respiratory functions of choir singers?
* Is diaphragmatic breathing exercise training provided by a physiotherapist effective in improving the vocal performance of choir singers?
* Does aerobic exercise training applied in addition to diaphragmatic breathing exercise training provided by a physiotherapist have a greater effect on improving the respiratory functions of choir singers compared to diaphragmatic breathing exercise training applied alone?
* Does aerobic exercise training applied in addition to diaphragmatic breathing exercise training provided by a physiotherapist have a greater effect on improving the vocal performance of choir singers compared to diaphragmatic breathing exercise training applied alone?

The research data are going to be collected by Sociodemographic Information Form, International Physical Activity Questionnaire-Short Form, Self-Performance Evaluation Questionnaire, Vocal Fatigue Index, Singing Voice Handicap Index, measurement of maximum phonation time, pulmonary function test, maximal inspiratory and expiratory pressure measurement, and 6-minute walk test.

DETAILED DESCRIPTION:
In this study, it will be examined whether aerobic exercise training applied in addition to diaphragmatic breathing exercise training provided by a physiotherapist improves respiratory functions and voice performance in choir singers more, when compared to diaphragmatic breathing exercise training applied alone.

The participants will be randomly divided into three groups: diaphragmatic breathing exercise training group, aerobic exercise training group applied in addition to diaphragmatic breathing exercise training, and control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a chorist in an active choir that rehearses at least once a week for an average of 2 hours
* Having an inactive or minimally active physical activity level according to the International Physical Activity Questionnaire-Short Form
* Being between the ages of 25-60
* Being willing to participate in the study

Exclusion Criteria:

* Having a neurological or orthopedic disease
* Having a condition related to the cardiopulmonary system that would prevent exercise according to the Physical Activity Readiness Questionnaire (PAR-Q)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
FEV1/FVC | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  Pulmonary function test with a spirometer will be performed on all participants to assess forced expiratory volume in 1 second and forced vital capacity.
Slow vital capacity | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  Pulmonary function test with a spirometer will be performed on all participants to assess slow vital capacity.
Maximal voluntary ventilation | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  Pulmonary function test with a spirometer will be performed on all participants to assess maximal voluntary ventilation.
Maximal inspiratory and expiratory pressure | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  An electronic respiratory pressure meter will be used to calculate maximal inspiratory and expiratory pressure
Maximum phonation time | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  Each participant will be asked to say the vowels "a, e, i, o, u" at their most comfortable pitch for as long as possible, and the time they can say them will be determined by a stopwatch.

SECONDARY OUTCOMES:
Aerobic capacity and endurance | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  6 Minute Walk Test will be performed on all participants to assess aerobic capacity and endurance.
Vocal fatigue | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  Vocal Fatigue Index which is a self-report questionnaire for identifying individuals with vocal fatigue and characterizing their complaints will be used to assess the vocal fatigue of all participants.
Singing voice and voice-related problems | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  Singing Voice Handicap Index will be used to assess the voice-related handicaps of all participants.
Voice performance | This outcome will be evaluated twice: before starting the exercise program and after implementing the exercise program for 8 weeks.
  The Self-Performance Evaluation Questionnaire, which is created by the researcher and is a scale in which the participant evaluates his/her own musical performance by scoring it between from 1 to 10, will be used to evaluate the performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Nur TUNALI VAN DEN BERG, Prof., Study Chair — İstanbul Medipol University; Sıla YILMAZ, PhD (c.), Principal Investigator — İstanbul Medipol University
Locations (1):
- Choric Culture Association, Istanbul, Turkey (Türkiye)